CLINICAL TRIAL: NCT06704191
Title: MC240502: Cancer CARE (Connected Access and Remote Expertise) Beyond Walls In-home iNtraVesIcal ThErapy (INVITE) Study - A Phase Ib/II, Single-Arm Trial of Delivering Intravesical Therapy for Bladder Cancer in Patients' Homes
Brief Title: In-home Intravesical Chemotherapy for the Treatment of Bladder Cancer, INVITE Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240502; UL1TR002377 (NIH); NCI-2024-09555 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-002176 (Other: Mayo Clinic Institutional Review Board); MC240502 (Other: Mayo Clinic)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Non-Muscle Invasive Bladder Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Cystoscopy; Docetaxel; Gemcitabine; Home Care Services; House Calls; Mitomycin; Mitozytrex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (BCG, gemcitabine, docetaxel, mitomycin) (Experimental): INDUCTION (PHASE IB COHORT AND PHASE II COHORT): Patients receive BCG intravesically over 1-2 hours, gemcitabine intravesically over 1-2 hours, gemcitabine intravesically over 1 hour followed by docetaxel intravesically over 1 hour or mitomycin C intravesically over 1-2 hours in the urology clinic. Treatment repeats once weekly in the home for up to 5 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE (PHASE II COHORT ONLY): Patients receive in-home BCG intravesically over 1-2 hours once weekly for 3 weeks, gemcitabine intravesically over 1-2 hours once monthly for 3 months, gemcitabine intravesically over 1 hour followed by docetaxel intravesically over 1 hour once monthly for 3 months or mitomycin C intravesically over 1-2 hours once monthly for 3 months in the absence of disease progression or unacceptable toxicity.
  Additionally, patients undergo cystoscopy at end of study and receive access to CCBW home health visits throughout the study.
  Interventions: Biological: BCG Solution; Procedure: Cystoscopy; Drug: Docetaxel; Drug: Gemcitabine; Other: Home Health Encounter; Drug: Mitomycin; Other: Questionnaire Administration

INTERVENTIONS:
Biological: BCG Solution — Given intravesically
  Other Names: Bacillus Calmette Guerin Solution; Bacillus Calmette-Guerin Solution; TICE BCG Solution
Procedure: Cystoscopy — Undergo cystoscopy
  Other Names: CS
Drug: Docetaxel — Given intravesically
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Gemcitabine — Given intravesically
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Other: Home Health Encounter — Receive access to CCBW home health visits
  Other Names: HH; Home; Home Care Visit; Home Health
Drug: Mitomycin — Given intravesically
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitomycin C; Mitomycin pyelocalyceal; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706; Mitolem
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase Ib/II trial compares the safety, tolerability and acceptability of intravesical chemotherapy given at home to in-clinic administration in patients with non-muscle invasive bladder cancer. Chemotherapy drugs, such as bacillus Calmette-Guerin (BCG), gemcitabine, docetaxel, and mitomycin C, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Standard of care chemotherapy for non-invasive bladder cancer is usually given directly into the bladder through a catheter (intravesical). This process requires numerous visits and can be disruptive to the lives of patients and caregivers. Bringing cancer care to the patients with in-home intravesical therapy may help reduce the disruption to daily lives. In-home intravesical chemotherapy may be safe and tolerable and may also be preferable to in-clinic administration in patients with non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety of in-home delivery of intravesical therapy. II. To assess the feasibility of in-home delivery of intravesical therapy.

SECONDARY OBJECTIVE:

I. To evaluate patient satisfaction with in-home intravesical therapy.

OTHER OBJECTIVES:

I. To assess patient-reported function and global health status/quality of life.

II. To assess patient-reported adverse events. III. To assess home days during study period. IV. To assess patient satisfaction with in-home intravesical therapy. V. To assess unplanned interactions with urological care team. VI. To describe disease-free survival rates following intervention period.

OUTLINE:

INDUCTION (PHASE IB COHORT AND PHASE II COHORT): Patients receive BCG intravesically over 1-2 hours, gemcitabine intravesically over 1-2 hours, gemcitabine intravesically over 1 hour followed by docetaxel intravesically over 1 hour or mitomycin (mitomycin C) intravesically over 1-2 hours in the urology clinic. Treatment repeats once weekly in the home for up to 5 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE (PHASE II COHORT ONLY): Patients receive in-home BCG intravesically over 1-2 hours once weekly for 3 weeks, gemcitabine intravesically over 1-2 hours once monthly for 3 months, gemcitabine intravesically over 1 hour followed by docetaxel intravesically over 1 hour once monthly for 3 months or mitomycin C intravesically over 1-2 hours once monthly for 3 months in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo cystoscopy at end of study and receive access to Cancer Care Beyond Walls (CCBW) home health visits throughout the study.

After completion of study treatment, patients are followed up at 12 weeks from registration and up to 1 year after registration.

ELIGIBILITY:
Inclusion Criteria:

* PHASE IB ONLY: Female or male patients with histologically confirmed non-muscle invasive bladder cancer (stage Ta, Tis, or T1) who are currently receiving induction therapy with one of the following eligible intravesical treatment regimens

  * Gemcitabine
  * Sequential gemcitabine/docetaxel
  * Bacillus Calmette-Guerin
  * Mitomycin C
* PHASE II ONLY: Female or male patients with histologically confirmed non-muscle invasive bladder cancer (stage Ta, Tis or T1) who are receiving maintenance therapy with an eligible regimen
* PHASE IB ONLY: Able to be successfully catheterized and able to tolerate first dost of intravesical therapy in the outpatient clinic
* Residing within the area serviced by supplier network
* Residence either has Wi-Fi or cellular data network connection for virtual telehealth visits
* Age ≥ 18 years at time of registration
* Signed informed consent form by patient
* Willing and able to comply with the study protocol in the investigator's judgment
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to follow birth control requirements for females and males of reproductive potential

Exclusion Criteria:

* Receiving any other investigational or standard of care agent which would be considered as a treatment for non-muscle invasive bladder cancer and is not part of the eligible treatment regimens
* Actively receiving any other treatment for cancer (except hormone therapy for breast or prostate cancer, or treatment for non-invasive skin cancer)
* Requiring 24/7 assistance with activities of daily living (ADLs)
* Current inpatient hospitalization (excluding admission to the Advanced Care at Home program)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Myocardial infarction ≤ 6 months
  * Wound healing disorder
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Anticipation of the need for major surgery during the course of study treatment
* Known allergy or previous intolerance to drug regimens
* Pregnancy or breastfeeding
* Hypersensitivity or allergy to polysorbate 80 or paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | 12 weeks
  The incidence, type, and severity of AEs experienced will be reported. The maximum grade for each type of AE will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Feasibility of in-home intravesical therapy | 12 weeks
  Feasibility will be indicated by the proportion of patients who receive at least 4 of 5 planned doses of induction therapy in the home within 12 weeks of the first dose of intravesical therapy (received in the outpatient clinic).

SECONDARY OUTCOMES:
Patient-preferred treatment location | Up to 1 year
  The frequency and proportion of patients who indicate a preference for in-home intravesical therapy versus a traditional setting will be assessed using the Patient Satisfaction and Feedback Questionnaire. The questionnaire consists of 4 questions related to receipt of care [answered on a 5-point scale (e.g., Excellent/Very Good/Good/Fair/Poor or Very Effective/Capable and Effective/Neutral/Somewhat Effective/Needs Development)]; 1 question related to preference for treatment location; 3 questions answered with yes, no, or uncertain; 1 question related to experience (better than expected, same as expected, worse than expected); and 1 opened ended for feedback as to what could have improved the experience.
Patient-reported likelihood to recommend at home therapy | Up to 1 year
  Will be assessed using the Patient Satisfaction and Feedback Questionnaire. The frequency and proportion of patients who would recommend in-home intravesical therapy to other patients will be reported. The questionnaire consists of 4 questions related to receipt of care [answered on a 5-point scale (e.g., Excellent/Very Good/Good/Fair/Poor or Very Effective/Capable and Effective/Neutral/Somewhat Effective/Needs Development)]; 1 question related to preference for treatment location; 3 questions related to acceptability and likely recommendation answered with yes, no, or uncertain; 1 question related to experience (better than expected, same as expected, worse than expected); and 1 opened ended for feedback as to what could have improved the experience.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D. Lyon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials